CLINICAL TRIAL: NCT00461019
Title: CardioFiT™ for Heart Failure - Safety and Efficacy Study Protocol
Brief Title: CardioFit™ for the Treatment of Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioControl Medical (Industry)
Responsible Party: Sponsor, BioControl Medical (B.C.M) Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-MS-01
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantation of the CardioFit system (Experimental)
  Interventions: Procedure: Implantation and activation of the vagus nerve stimulator

INTERVENTIONS:
Procedure: Implantation and activation of the vagus nerve stimulator — Implantation of the nerve stimulator, cuff nerve electrode and RV sensing lead

SUMMARY:
Congestive Heart Failure is the result of a number of diseases affecting the heart, causing the heart's failure to properly meet the body demands for blood circulation. In spite of advances in drug therapy, it remains a significant public health problem.

Pharmacologic antagonism of the beta-adrenergic receptors shifting the autonomic balance in the direction of greater vagal influence is a well-proven treatment for heart failure patients, although there are patients who cannot tolerate, or only partially benefit from such a treatment.

It has been proven in the past and well established that parasympathetic nerve stimulation can slow the rate of the heart and reduce the workload of the heart. Therefore, the potential benefit of vagus nerve stimulation, hence parasympathetic activation, for treatment of heart failure is substantial.

In this study, the safety and efficacy of a new vagus nerve stimulating system will be evaluated. This study will compare whether the new device improves Heart Failure parameters in Class II - III Heart Failure patients.

DETAILED DESCRIPTION:
* Purpose of the study: To determine the safety and efficacy of the CardioFit™ system for treatment of Class II-III Heart Failure patients.
* Study hypothesis: CardioFit system treatment will improve patients Heart Failure parameters.
* Tested hypothesis: Thirty patients are required to provide 80% power at 95% confidence level in order to detect 12 points difference on a quality of life questionnaire between pre- and post activation.
* Design: Prospective, self-controlled interventional study composed of 5 periods: Pre-implantation, Implantation, Device activation, Follow-up (with active device) and post-study extension period.
* Study duration is 7.5-months per patient. At the end of the study, patients enter an extension period (with active devices) during which they will be monitored for quality of life and survival, for up to 3 years post-implantation in 6-months intervals.
* Study Endpoints:

  * Primary endpoints: The occurrence of all system and/or procedure related adverse events.
  * Secondary endpoints: changes in the following individual variables as well as in a composite score of individual variables change: NYHA class; Quality of Life; Exercise capacity (by 6-min walk); LV Ejection fraction; LV end-systolic and end-diastolic volumes; blood tests.
* Up to 10 participating centers in Europe, Israel and Australia

ELIGIBILITY:
Inclusion Criteria:

1. The patient is in chronic heart failure, NYHA II-III. The patient may have been previously in class IV but must be in class II or III for three or more months prior to study entry;
2. Age between 18 and 75 years;
3. The patient is a male or postmenopausal female. Females of childbearing age may be included if pregnancy is excluded and acceptable contraception measures are used;
4. Patient must sign an approved informed consent form. Patient agrees to attend all follow-up evaluations;
5. Patient should be in sinus rhythm. Average 24-hour heart rate is between 60 and 110 b/min in a recorded 24-h Holter measurement;
6. Patient should be in optimal medical treatment with no change in treatment in the previous 3 months with the exception of diuretics;
7. Left ventricular ejection fraction estimated by echocardiography, cardiac angiography, radionuclide study, or other accepted mode of evaluation, is no more than 35%;
8. Patient is physically capable and willing to perform repeated physically demanding tests associated with the study.

Exclusion Criteria:

1. Presence of an immediately life threatening condition or disease other than heart failure, such as cancer, terminal renal failure etc.
2. Acute myocardial Infarction (MI), variant angina pectoris, unstable angina or acute coronary syndrome in the previous three months;
3. Previous stroke;
4. Coronary Artery Bypass Surgery (CABG) or Percutaneous Coronary Intervention in the past 3 months;
5. Episode of NYHA class IV heart failure, including acute pulmonary oedema in the previous three months;
6. Heart failure due to acute myocarditis. Restrictive or constrictive pericarditis, haemodynamically significant aortic valve insufficiency aortic stenosis, or mitral valve stenosis;
7. Severe renal or hepatic failure (Creatinine level>3 mg% (265 micromole/liter) or transaminase level four times ULN);
8. Diabetes Mellitus treated with insulin for more than two years prior to study entry;
9. Diabetic neuropathy;
10. Previous neck surgery, including for Peripheral Vascular Disease (PVD), malignancy, and previous irradiation therapy of the neck;
11. Current hypotension (systolic blood pressure below 80 mmHg);
12. Active peptic disease or history of upper GI bleeding;
13. Asthma, severe COPD (e.g. FEV1<1.5 liter), or severe restrictive lung disease;
14. 1st degree AV block with PR interval > 240msec, 2nd or 3rd degree AV block;
15. Atrial fibrillation or flutter in the in the previous 3 months;
16. Sustained ventricular tachyarrhythmia with hemodynamic compromise, in the absence of implanted ICD;
17. Long QT syndrome, congenital or acquired;
18. Recorded or suspected symptomatic vaso-vagal response;
19. Treatment by investigational drug or device within the past 3 months;
20. Glaucoma, or history of glaucoma;
21. Major psychiatric disorder in the present or in the past; Dementia;
22. Patients transplanted with tissues or organs;
23. Immunosuppressed patients; patients under systemic steroid treatment;
24. Anemia with Hb<10gr/L, unless treated with Epo;
25. Patients who are at risk for carotid arteries plaques and have unstable carotid plaques, as assessed by Echo Doppler; and/or patients with >70% carotid artery stenosis;
26. Patient is candidate for cardiac resynchronization device implantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The occurrence of all system and/or procedure related adverse events. | along the study

SECONDARY OUTCOMES:
Change in NYHA class | At 6-months
Quality of Life | At 6-months
Exercise capacity (by 6-min walk) | At 6-months
LV Ejection fraction | At 6-months
LV end-systolic and end-diastolic volumes | At 6-months
Blood tests. | At 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schwartz, Professor, Principal Investigator — Fondazione IRCCS Policlinico San-Matteo
Locations (6):
- Germany (3):
  - Georg-August-Universität Göttingen, Göttingen
  - Otto von-Guericke University Clinik, Magdeburg
  - I. Medizinische Klinik, Klinikum Mannheim GmbH Universitätsklinikum Fakultät für klinische Medizin Mannheim der Universität Heidelberg, Mannheim
- Fondazione IRCCS Policlinico "San Matteo", Pavia, Pavia, Italy
- Academic Hospital Maastricht, Maastricht, Netherlands
- Pacemaker center, Cardiovascular institute Clinical Center of Serbia, Belgrade, Serbia

REFERENCES:
- [Result] De Ferrari GM, Crijns HJ, Borggrefe M, Milasinovic G, Smid J, Zabel M, Gavazzi A, Sanzo A, Dennert R, Kuschyk J, Raspopovic S, Klein H, Swedberg K, Schwartz PJ; CardioFit Multicenter Trial Investigators. Chronic vagus nerve stimulation: a new and promising therapeutic approach for chronic heart failure. Eur Heart J. 2011 Apr;32(7):847-55. doi: 10.1093/eurheartj/ehq391. Epub 2010 Oct 28. PMID 21030409
- [Result] Schwartz PJ, De Ferrari GM, Sanzo A, Landolina M, Rordorf R, Raineri C, Campana C, Revera M, Ajmone-Marsan N, Tavazzi L, Odero A. Long term vagal stimulation in patients with advanced heart failure: first experience in man. Eur J Heart Fail. 2008 Sep;10(9):884-91. doi: 10.1016/j.ejheart.2008.07.016. Epub 2008 Aug 28. PMID 18760668
- See also: INOVATE-HF INcrease Of VAgal TonE in Heart Failure — http://www.clinicaltrials.gov/ct2/show/NCT01303718?term=BioControl+Medical&rank=1